CLINICAL TRIAL: NCT00982917
Title: Stamp-in-Safety Playground Safety Project
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Collaborators: Robert Wood Johnson Foundation (Other); Kohl's Cares for Kids Safety Network (Unknown)
Responsible Party: Karen Sheehan, MD, MPH, Children's Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2006-12867
Record Dates: First submitted 2009-09-22; First posted 2009-09-23 (Estimated); Last update posted 2009-09-23 (Estimated); Status verified 2009-09

CONDITIONS: Injury Prevention
Keywords: playground; injury prevention

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- teachers taught curriculum (Experimental): Teachers taught Stamp-in-Safety curriculum
  Interventions: Behavioral: Stamp-in-Safety Curriculum
- teachers do not learn curriculum (Experimental): Teachers are not taught Stamp-in-Safety curriculum
  Interventions: Behavioral: Stamp-in-Safety Curriculum

INTERVENTIONS:
Behavioral: Stamp-in-Safety Curriculum — 30 minute curriculum on playground safety
Behavioral: Stamp-in-Safety curriculum — 30 minute lesson on playground supervision

SUMMARY:
Playground injuries are common at childcare centers. Adequate adult supervision is an important component to reducing playground injuries in preschool children. The investigators studied the Stamp-in-Safety Program, an intervention to improve adult supervision and reduce children's risky playground behaviors.

DETAILED DESCRIPTION:
Using a non-equivalent control group design, we evaluated the Stamp-in-Safety program which increases the quality of adult supervision and rewards children for safe play. In an urban childcare center, 71 children, ages 3-5 years, and 15 teachers participated in the study. The primary outcome measures were teacher verbalizations (warnings, explanations, redirects), teacher location (core, outskirts, or fringe of playground), risk taking behaviors by children (using equipment appropriately), and number of injuries on the playground.

ELIGIBILITY:
Inclusion Criteria:

* teachers at childcare center
* students at childcare center

Exclusion Criteria:

* not affiliated with childcare center

Ages: 3 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 71 (Actual)
Dates: Start 2006-06; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
Improve adult supervision on playgrounds | 5 weeks

SECONDARY OUTCOMES:
Decrease preschool children's risky behaviors on playgrounds | 5 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Karen Sheehan, MD, MPH, Principal Investigator — Ann & Robert H Lurie Children's Hospital of Chicago
Locations (1):
- ST. Vincent De Paul Childcare Center, Chicago, Illinois, United States